CLINICAL TRIAL: NCT02989662
Title: Glucocorticoid Antagonists in Heavy Drinkers: Effects on fMRI Connectivity, Withdrawal and Drinking
Brief Title: INIA Stress and Chronic Alcohol Interactions: Glucocorticoid Antagonists in Heavy Drinkers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00138426; U01AA020890 (NIH); AA020890 (Other: Other)
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Alcohol Use Disorder - Mifepristone (Active Comparator): Participants diagnosed with alcohol use disorder who were randomized to receive mifepristone. Mifepristone is a high affinity antagonist of the glucocorticoid receptor (GR). It is FDA approved to treatment hyperglycemia caused by high cortisol levels in adults with endogenous Cushing's syndrome.
  Interventions: Drug: Mifepristone
- Alcohol Use Disorder - Placebo (Placebo Comparator): Participants diagnosed with alcohol use disorder who were randomized to receive placebo. This is an inactive compound which appears physically identical to active medication.
  Interventions: Drug: Placebo - Cap
- Healthy Control - Mifepristone (Active Comparator): Healthy control participants who were randomized to receive mifepristone. Mifepristone is a high affinity antagonist of the glucocorticoid receptor (GR). It is FDA approved to treatment hyperglycemia caused by high cortisol levels in adults with endogenous Cushing's syndrome.
  Interventions: Drug: Mifepristone
- Healthy Control - Placebo (Placebo Comparator): Healthy control participants who were randomized to receive placebo. This is an inactive compound which appears physically identical to active medication.
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Mifepristone — Participants receive 6 doses.
  Other Names: Korlym
  Arms: Alcohol Use Disorder - Mifepristone; Healthy Control - Mifepristone
Drug: Placebo - Cap — Participants receive 6 doses
  Arms: Alcohol Use Disorder - Placebo; Healthy Control - Placebo

SUMMARY:
In alcohol use disorder (AUD) and matched healthy control (HC) men and women, the proposed research examines the effects of MIFE, with demonstrated preclinical effects on drinking-related behaviors, compared with placebo on a breadth of alcohol-related measures. All subjects will be randomized to daily MIFE or placebo. Before and during medication, AUD and HC subjects undergo fMRI scanning measuring resting-state functional connectivity and alcohol cue-induced brain activation focused on brain reward and stress pathways. All subjects are admitted to the Clinical Research Unit; AUD subjects undergo supervised alcohol withdrawal with daily measurements of alcohol craving and symptom severity. Using validated human laboratory procedures in AUD subjects, this study will examine the effects of stress on motivation to drink and alcohol sensitivity/reward as a function of GR antagonism.

DETAILED DESCRIPTION:
Cortisol (CORT) is a glucocorticoid hormone, often associated with response to stress and playing a key role in alcohol use and problems. First, acute alcohol administration increases CORT, which in turn amplifies the mesolimbic dopamine reward signal. Second, alcohol withdrawal elevates CORT levels in AUD compared with healthy control subjects, and CORT levels in early abstinence predict subsequent relapse to drinking. Finally, the magnitude of CORT response to external stressors predicts motivation to work for and consumption of alcohol in the human laboratory and in the natural environment. Importantly, recent studies in rodents and humans have demonstrated that blocking CORT activity using a glucocorticoid receptor (GR) antagonist reduces these effects of CORT on alcohol behaviors, indicating a causal role for glucocorticoids in these relationships. In alcohol use disorder (AUD) and matched healthy control (HC) men and women, the proposed research examines the effects of MIFE, with demonstrated preclinical effects on drinking-related behaviors, compared to placebo on a breadth of alcohol-related measures. All subjects will be randomized to daily MIFE or placebo. Before and during medication, AUD and HC subjects undergo fMRI scanning measuring resting-state functional connectivity and alcohol cue-induced brain activation focused on brain reward and stress pathways. All subjects are admitted to the Clinical Research Unit; AUD subjects undergo supervised alcohol withdrawal with daily measurements of alcohol craving and symptom severity. Using validated human laboratory procedures in AUD subjects, this study will examine the effects of stress on motivation to drink and alcohol sensitivity/reward as a function of GR antagonism. This work will help pave the way for improved pharmacotherapies that target stress and reward pathways in the brain involved in initiating and maintaining drinking.

ELIGIBILITY:
Inclusion Criteria:

* Nontreatment seeking AUD volunteers
* English speaking
* healthy
* Not pregnant or nursing

Exclusion Criteria:

* Women on hormonal birth control, pregnant or nursing
* Current health or psychiatric problems
* Potassium level below normal
* Any medication or health condition that is known to interact with MIFE or CORT metabolism
* History of metal implantation that would preclude MRI scan.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E McCaul, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Integrated Program for Substance Abuse Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 65 participants who were consented for the study, 33 were determined to be ineligible during the assessment procedures. Among the 32 persons who were eligible, 16 were not randomized to study medication (8 participants were lost to follow-up and 8 participants withdrew from the study).
Period: Overall Study
Arm/Group | Alcohol Use Disorder - Mifepristone | Alcohol Use Disorder - Placebo | Healthy Control - Mifepristone | Healthy Control - Placebo
Started (Completed baseline assessment, determined to be study eligible and randomized to study medication condition.) | 4 | 3 | 6 | 3
Completed | 0 | 3 | 6 | 1
Not Completed | 4 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Physician Decision | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol Use Disorder - Mifepristone | Alcohol Use Disorder - Placebo | Healthy Control - Mifepristone | Healthy Control - Placebo | Total
Number analyzed (Participants) | 4 | 3 | 6 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.8) | 41.3 (7.1) | 38.3 (13.8) | 33.7 (8.6) | 39.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 0 | 4
  Male | 3 | 1 | 5 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 2 | 8
  White | 1 | 1 | 3 | 1 | 6
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 6 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Oxygen Level Dependent (BOLD) fMRI Signal for Alcohol Versus Non-alcohol Stimuli
Description: Participants observed alcohol and neutral cues during functional MRI (fMRI) scans. Larger numbers indicate greater activation to alcohol versus non alcohol stimuli. Mean response Pre and Post medication (mifepristone (MIFE), placebo), is measured. The greater the number the greater the reactivity to alcohol-related cues.
Time Frame: Change from baseline (Day 1) to day 4 of MIFE dosing
Population: No data were collected for the AUD Mifepristone participants. AUD Mifepristone participants either dropped out or were withdrawn from the study prior to fMRI procedures. In addition, fMRI data were lost on one AUD-Placebo participant and one Healthy Control - Placebo participant due to head movement artifact.
Measure: Mean (Standard Error); unit: BOLD response
Arm/Group | Alcohol Use Disorder - Mifepristone | Alcohol Use Disorder - Placebo | Healthy Control - Mifepristone | Healthy Control - Placebo
Number analyzed (Participants) | 0 | 2 | 6 | 2
BOLD response
  Amygdala, centromedian - day 1 |  | 0.267390 (0.128827) | 0.040281 (0.074378) | 0.058670 (0.128827)
  Amygdala, centromedian - day 4 |  | -0.069048 (0.142952) | 0.037178 (0.082533) | 0.052388 (0.142952)
  Amygdala, lateral - day 1 |  | 0.091174 (0.190861) | 0.151864 (0.110194) | 0.099169 (0.190861)
  Amygdala, lateral - day 4 |  | 0.294417 (0.115607) | -0.021411 (0.066746) | 0.126445 (0.115607)
  medial prefrontal cortex - day 1 |  | 0.044635 (0.287281) | -0.323039 (0.165862) | 0.031454 (0.287281)
  medial prefrontal cortex - day 4 |  | 0.439822 (0.226576) | 0.257514 (0.130814) | -0.514729 (0.226576)
  nucleus accumbens - day 1 |  | 0.138441 (0.147427) | 0.131360 (0.085117) | 0.262425 (0.147427)
  nucleus accumbens - day 4 |  | 0.285409 (0.106153) | 0.138914 (0.061287) | -0.003538 (0.106153)
  Amygdala, superficial - day 1 |  | 0.583073 (0.269851) | 0.252555 (0.155799) | -0.111622 (0.269851)
  Amygdala, superficial - day 4 |  | 0.149175 (0.347008) | 0.172212 (0.200345) | 0.118748 (0.347008)
  ventral tegmental area - day 1 |  | 0.405165 (0.227379) | 0.566876 (0.131277) | -0.019192 (0.227379)
  ventral tegmental area - day 4 |  | 0.430387 (0.176868) | -0.150802 (0.102115) | 0.104408 (0.176868)

2. Secondary Outcome: Mean of Alcohol Motivated Responses Made
Description: Participants made alcohol motivated responses with a computer mouse to earn either alcohol drinks or money. Each mouse click equaled one response. Mean of all responses made are reported.
Time Frame: single session on study day 5
Population: This measure was designed to only be collected among the participants with alcohol use disorder (AUD). None of the AUD participants randomized to mifepristone completed the study. No data were collected for AUD-Mifepristone participants as they either dropped out or were withdrawn from the study prior to completing this procedure.
Measure: Mean (Standard Deviation); unit: responses made
Groups:
- Healthy Control - Mifepristone: Healthy control participants who were randomized to receive mifepristone. Mifepristone is a high affinity antagonist of the glucocorticoid receptor (GR). It is FDA approved to treatment hyperglycemia caused by high cortisol levels in adults with endogenous Cushing's syndrome.
  Healthy controls did not participate in this study procedure.
- Healthy Control - Placebo: Healthy control participants who were randomized to receive placebo. This is an inactive compound which appears physically identical to active medication.
  Healthy controls did not participate in this study procedure.
Arm/Group | Alcohol Use Disorder - Mifepristone | Alcohol Use Disorder - Placebo | Healthy Control - Mifepristone | Healthy Control - Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 0
responses made |  | 9517 (1497.6) |  |

3. Secondary Outcome: Alcohol Motivated Responding - Number of Drinks Earned
Description: Participants can earn up to 10 drinks during a 1-hr session. Each drink was the equivalent of 0.5 standard drink.
Time Frame: single session on study day 5
Population: This measure was designed to only be collected among the participants with alcohol use disorder (AUD). None of the AUD participants randomized to mifepristone completed the study. No data were collected for participants in the AUD-Mifepristone group. Participants either dropped out or were withdrawn from the study before completing this procedure.
Measure: Mean (Standard Deviation); unit: drinks earned
Arm/Group | Alcohol Use Disorder - Mifepristone | Alcohol Use Disorder - Placebo | Healthy Control - Mifepristone | Healthy Control - Placebo
Number analyzed (Participants) | 0 | 3 | 0 | 0
drinks earned |  | 7 (3) |  |

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post followup
Groups:
- Health Control - Placebo: Healthy control participants who were randomized to receive placebo. This is an inactive compound which appears physically identical to active medication.
Arm/Group | Alcohol Use Disorder - Mifepristone | Alcohol Use Disorder - Placebo | Healthy Control - Mifepristone | Health Control - Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 2/6 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcohol Use Disorder - Mifepristone (N=4) | Alcohol Use Disorder - Placebo (N=3) | Healthy Control - Mifepristone (N=6) | Health Control - Placebo (N=3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT02989662/Prot_SAP_000.pdf